CLINICAL TRIAL: NCT06192628
Title: A Randomised Controlled Feasibility Study to Promote Physical Activity and Exercise Adherence Among People With Parkinson's
Brief Title: Behavioural Change Techniques for Physical Activity and Exercise Adherence Among People With Parkinson's
Acronym: PDActive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Ruth McCullagh, Lecturer in Physiotherapy, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20114
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
Keywords: behavioural change intervention; exercise self-efficacy; exercise adherence; physiotherapy; theoretical domains framework
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: two-arm single blinded randomised feasibility study
Who Masked: Participant
Masking Description: patients are randomly allocated using concealed envelopes, and they are not informed as to which arm they have been allocated. They both receive an exercise programme, with the active arm receiving additional behavioral change techniques to promote exercise adherence and exercise self efficacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's Education and Exercise Programme [PEEP] (Active Comparator): 12 week programme of exercises and educational sessions
  Interventions: Behavioral: Parkinson's Exercise and Education Programme
- Parkinson's Education and Exercise Programme and Behavioural Change [PEEP-BC] (Experimental): 12 week programme of exercise and education with additional behavioural change techniques to promote exercise adherence and exercise self-efficacy.
  Interventions: Behavioral: Parkinson's Exercise and Education Programme and Behavioural Change

INTERVENTIONS:
Behavioral: Parkinson's Exercise and Education Programme — A 12 week programme of exercise and education
  The weekly programme consists of a 45-minute exercise programme, 45-minute education sessions delivered by healthcare professionals about their role in Parkinson's management, and independent home exercise programmes completed twice weekly (determined by the registered physiotherapist only)
  Arms: Parkinson's Education and Exercise Programme [PEEP]
Behavioral: Parkinson's Exercise and Education Programme and Behavioural Change — A 12-week programme of exercise, education and behavioural change techniques to support exercise adherence and exercise self-efficacy
  The weekly programme consists of a 45-minute exercise programme, 45-minute education sessions delivered by healthcare professionals about their role in Parkinson's management, and independent home exercise programmes completed twice weekly (determined by the registered physiotherapist and participant)
  Additional techniques addressing behavioural regulation include firstly, an exercise diary completed independently at home, secondly, the rationale and the intended functional benefit and expectations of the exercise programme clearly explained, thirdly individual weekly conversations to reflect on progress, expectations, solutions to barriers, and goals. Finally, peer support is strongly encouraged through the in-class support, and a social media networking group.
  Arms: Parkinson's Education and Exercise Programme and Behavioural Change [PEEP-BC]

SUMMARY:
Many people with Parkinson's (PwP) experience many barriers to reaching the recommended dosage of exercise. The aim of this study is to examine the feasibility of behavioural change support techniques delivered alongside an exercise programme to improve physical activity, function, to inform a future pilot randomised controlled trial.

Twenty participants with Parkinson's will be allocated to the intervention (n=10) or the control group (n=10). Both groups will receive usual care, which includes a weekly program of a multidisciplinary education, a supervised exercise class and a prescribed home exercise program. The intervention group will receive additional behavioural change techniques to help them adhere to the exercises, targeting behaviour regulation, belief about capabilities and social influences.

Outcomes will measure how well people were able to stay in the programme, and their physical function after the 12 week programme. Surveys will be used to compare experiences and satisfaction between groups. Exit interviews will be completed with the intervention group only, exploring their experience of the behavioural change techniques.

Discussion: The results will help inform a future pilot randomised controlled trial, based on the intervention acceptability, consent rate, maintenance, and protocol integrity.

DETAILED DESCRIPTION:
Background: Parkinson's is a common progressive neurological condition characterized by motor and non-motor deficits. Physical activity and exercise can improve health, but many people with Parkinson's (PwP) have trouble reaching the recommended dosage. Our recent literature review found improvements in exercise adherence with behavioural change interventions, but it remains unclear which are most effective. Further qualitative research and patient and public involvement has informed a novel behavioural change support intervention to be tested alongside an existing exercise program.

Objective: To examine the feasibility of behavioural change support techniques delivered alongside an exercise programme to improve physical activity, function, and self-efficacy in PwP (and study procedures) to inform a future pilot RCT trial.

Methods: A parallel-arm single blinded randomised feasibility study. Twenty participants with Parkinson's (Hoehn and Yahr stage 1-3) will be recruited from a physiotherapy primary-care waiting list. Following written consent, and baseline assessment, the participants will be randomly allocated to the intervention (n=10) or the control group (n=10). Both groups will receive usual care, which includes a weekly program of a multidisciplinary education, a supervised exercise class and a prescribed home exercise program. The intervention group will receive additional behavioural change techniques, targeting behaviour regulation, belief about capabilities and social influences. Class and home exercise adherence, behavioural component uptake and adherence, and negative events will be recorded. Outcomes will include enrolment and maintenance rates, physical function, falls, physical activity, and exercise self-efficacy measured pre- and post- the 12- week program (in-person). Surveys will be used to compare experiences and satisfaction between groups. Exit interviews will be completed with the intervention group only, exploring their experience of the behavioural change techniques.

Discussion: The results will help inform a future pilot RCT, based on the intervention acceptability, consent rate, maintenance, and protocol integrity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease (Early Stages of Parkinson's H&Y Stage 1-3)
* Ability to drive or obtain transport that will drop and collect at the health centre.
* Ability to independently walk (with or without a walking aid)
* Reported by the referring healthcare provider or carer as able to follow instructions and carry out the exercise program independently at home.

Exclusion Criteria:

* • A diagnosis of atypical Parkinson's (e.g., progressive supranuclear palsy, multiple system atrophy, etc) or vascular Parkinsonism or drug-induced parkinsonism

  * Previously completed the PEEP program.
  * Had a hospital admission < 6 weeks ago.
  * Immobility, or are a wheelchair-user.
  * Severe visual or auditory impairment
  * Serious medical conditions in major organs (heart, lung, or kidney) or other illnesses which prevent independent ambulation or safe exercise.
  * Been identified as a high falls risk (identified during the pre-screening using objective measure the Short Physical Performance Battery (a score of ≤6 indicates a higher fall risk in old adults27) and subjective reporting of frequent falls in the past six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Average daily step-count | week 0 and week 12
  Accelerometry data measuring one week of walking
Incidence of falls in the previous three months (self-reported) | week 0 and week 12
  recorded falls and near falls events
Timed Up and Go Test (Walking speed; metres per second) | week 0 and week 12
  APDM Mobility Lab sensor-based gait and balance analysis system to objectively measure Timed Up and Go test and a 2-minute free walking test
Two Minute Free Walking Test (Walking Speed; metres per second) | week 0 and week 12
  APDM Mobility Lab sensor-based gait and balance analysis system to objectively measure Timed Up and Go test and a 2-minute free walking test
Exercise Self-efficacy Scale | week 0 and week 12
  [Self reported] Exercise Self Efficacy Scale, validated in people with Parkinson's (score range 10-40, higher indicating more confidence.)

SECONDARY OUTCOMES:
Exercise endurance | week 0 and week 12
  Six minute walk test
Health related Quality of Life | week 0 and week 12
  Parkinson's Disease Questionnaire-39 (PDQ-39). The scale contains 39 items covering eight dimensions of health status. Possible scores range between 0-100, with lower scores reflect better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth McCullagh, PhD, Principal Investigator — University College Cork
Locations (1):
- St Marys Primary Care Centre, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Yes
We plan to share aggregated data and store anonymised data on an open repository linked to the published report of the study, with a unique digital object identifier (DOI).
Supporting Information: Study Protocol, ICF
Time Frame: June 2024, with no time limit
Access Criteria: unknown as yet

REFERENCES:
- [Derived] Ahern L, Timmons S, Lamb SE, McCullagh R. Behaviour Change for Parkinson's Disease: A Randomised Controlled Feasibility Study to Promote Physical Activity and Exercise Adherence Among People with Parkinson's Disease. J Frailty Sarcopenia Falls. 2025 Sep 1;10(3):128-149. doi: 10.22540/JFSF-10-128. eCollection 2025 Sep. PMID 40901341
- [Derived] Ahern L, Timmons S, Lamb SE, McCullagh R. Behavioural change for Parkinson's Disease: A randomised controlled feasibility study to promote physical activity and exercise adherence among people with Parkinson's: study protocol. HRB Open Res. 2024 May 29;7:7. doi: 10.12688/hrbopenres.13843.2. eCollection 2024. PMID 38784965